CLINICAL TRIAL: NCT07067645
Title: Investigation of the Effect of Horizontal and Vertical Vaginal Cuff Closure on Postoperative Total Vaginal Length in Patients Undergoing Vaginal Hysterectomy and Lateral Suspension
Brief Title: Post-Hysterectomy Vaginal Length: Horizontal vs. Vertical Closure
Acronym: vagina
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Serkan Kumbasar, Associate Professor, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gopvaginallength
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Prolapse, Vaginal; Vaginal Vault Prolapse
Keywords: Vault suspension; vaginal length
MeSH Terms: conditions — Uterine Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel-assignment clinical study designed to compare two surgical techniques for vaginal cuff closure-horizontal versus vertical-performed during vaginal hysterectomy with lateral suspension for uterine prolapse. Patients will be randomly assigned to one of two intervention arms, with the aim of evaluating the impact of closure orientation on total postoperative vaginal length. The study will be conducted at a single center with standardized surgical and measurement protocols, and outcomes will be assessed by blinded evaluators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horizontal Vaginal Cuff Closure (Active Comparator): Patients in this group will undergo vaginal hysterectomy with lateral suspension, followed by horizontal closure of the vaginal cuff using standard suturing technique. The effect on postoperative total vaginal length will be evaluated.
  Interventions: Procedure: Horizontal Vaginal Cuff Closure Technique
- Vertical Vaginal Cuff Closure (Active Comparator): Patients in this group will undergo vaginal hysterectomy with lateral suspension, followed by vertical closure of the vaginal cuff using standard suturing technique. Postoperative vaginal length outcomes will be compared to those of the horizontal closure group.
  Interventions: Procedure: Vertical Vaginal Cuff Closure Technique

INTERVENTIONS:
Procedure: Horizontal Vaginal Cuff Closure Technique — In this arm, patients undergoing vaginal hysterectomy with lateral suspension will receive horizontal closure of the vaginal cuff. After removal of the uterus, the vaginal cuff is closed in a transverse (right-to-left) direction using standard absorbable sutures. The technique aims to maintain or optimize the anatomical axis and preserve vaginal length in the horizontal plane. The entire procedure is performed under general or regional anesthesia by an experienced surgical team.
  Arms: Horizontal Vaginal Cuff Closure
Procedure: Vertical Vaginal Cuff Closure Technique — In this arm, patients undergoing vaginal hysterectomy with lateral suspension will receive vertical closure of the vaginal cuff. After the uterus is removed, the vaginal cuff is closed in a cranio-caudal (top-to-bottom) orientation using absorbable sutures. This technique is hypothesized to better support apical structures and reduce tissue tension. Procedures are performed under general or regional anesthesia with standardized operative technique.
  Arms: Vertical Vaginal Cuff Closure

SUMMARY:
This prospective clinical study aims to evaluate the impact of vaginal cuff closure orientation-horizontal versus vertical-on postoperative total vaginal length in patients undergoing vaginal hysterectomy combined with lateral suspension. By comparing anatomical outcomes between the two closure techniques, the study seeks to determine which method better preserves vaginal length, potentially influencing surgical preferences and postoperative quality of life.

DETAILED DESCRIPTION:
This prospective clinical study is designed to evaluate the effect of vaginal cuff closure orientation-horizontal versus vertical-on postoperative total vaginal length in patients undergoing vaginal hysterectomy with lateral suspension. Vaginal length is a significant factor in pelvic floor support, sexual function, and patient satisfaction after pelvic organ prolapse surgeries.

Eligible patients undergoing vaginal hysterectomy and lateral suspension for uterine prolapse will be randomly assigned to two groups based on the vaginal cuff closure technique: Group 1 (horizontal closure) and Group 2 (vertical closure). All surgeries will be performed by the same surgical team to minimize technique-related variability. Preoperative and postoperative total vaginal lengths will be measured via standardized pelvic examination and recorded.

Secondary outcomes will include patient-reported symptoms (e.g., sensation of vaginal shortening, sexual function), surgical duration, intraoperative complications, and early postoperative outcomes. The study aims to provide evidence-based guidance on optimal vaginal cuff closure technique in uterovaginal prolapse surgery, with an emphasis on preserving vaginal length and improving postoperative quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cases with vaginal hysterectomy and lateral suspension surgery due to stage 3-4 uterine prolapse Agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* Cases that have previously undergone a different suspension surgery due to descent uteri (vaginal hysterectomy and sacrospinous ligament fixation surgery, vaginal hysterectomy and sacrocolopexy surgery, vaginal hysterectomy and high sacouterin plication surgery) Cases that have undergone vaginal hysterectomy due to malignancy Cases that have undergone radiotherapy due to malignancy (brachytherapy) Patients who are not suitable for surgical intervention due to severe vaginal atrophy.

Patients who will not be able to comply with the follow-up process. Not accepting to participate in the study or not signing the informed consent form

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POP-Q) Score | Baseline, 3 and 6 months postoperatively
  POP-Q scores will be used to assess anatomical outcomes of the pelvic support structures before and after surgery. Standardized POP-Q measurements (Aa, Ba, C, D, Ap, Bp, gh, pb, tvl) will be recorded preoperatively, 3 and 6 months postoperatively by blinded examiners. The primary focus will be on point C (vaginal apex) and total vaginal length (TVL) for comparison between groups.
PISQ-12 Questionnaire Score | Baseline, 3 and 6 months postoperatively
  The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) will be administered to sexually active patients preoperatively, 3 and 6 months postoperatively to assess sexual function and satisfaction. Changes in the total PISQ-12 score will be analyzed between the horizontal and vertical closure groups.

CONTACTS AND LOCATIONS:
Overall Officials: yagmur acıyiyen, md, Principal Investigator — Gaziosmanpasa Training and Research Hospital
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No